CLINICAL TRIAL: NCT06353672
Title: A Study to Evaluate Safety and Feasibility of Robotic Liver Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RLR-01
Record Dates: First submitted 2024-03-26; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Liver Diseases; Surgery
Keywords: Robotic liver resection
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic liver resection (Experimental)
  Interventions: Device: Robotic liver resection

INTERVENTIONS:
Device: Robotic liver resection — Liver resection using Da Vinci robotic system

SUMMARY:
The robotic surgery system, the most advanced technology in minimally invasive surgery, overcame some shortcomings of laparoscopic surgery and improved the flexibility and precision of liver resection. Several studies have demonstrated that the robotic system was safe and feasible in liver surgery and might be advantageous in complex hepatic vein and hilar dissection, operative bleeding control, and biliary reconstruction. Previous comparative studies found limited evidence for significantly improved outcomes in robotic liver resection (RLR) over laparoscopic liver resection (LLR) or open liver resection (OLR), considering the various degrees of difficulty in liver surgeries.

This study aimed to evaluate safety and feasibility of robotic liver resection, by comparing it with LLR or OLR, and gain veritable and relevant data on the benefits of RLR.

ELIGIBILITY:
Inclusion Criteria:

* The patients were diagnosed with a liver tumor.
* The patients underwent robotic liver resection.

Exclusion Criteria:

* The patients underwent simultaneous malignancy resection of the colorectum or other organs (except gallbladder).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | with in 90 days after surgery
  The grades of postoperative complications were recorded following the Clavien-Dindo classification. Partial hepatic dysfunction or hepatic failure, biliary fistula, postoperative hemorrhage, pleural effusion, venous thrombosis, and surgical site infections were recorded.
Postoperative hospital stay | with in 90 days after surgery
  The days of hospital stay after operation
Postoperative unplanned reoperation | with in 90 days after surgery
  The unplanned reoperation due to postoperative complications
Unplanned readmission | with in 90 days after surgery
  The unplanned readmission after discharge due to postoperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Medical College of Zhejiang University, Hangzhou, Zhejiang, China